CLINICAL TRIAL: NCT01244880
Title: Subject And Investigator-Blinded, Sponsor-Open, Randomized, Single-Dose, Placebo-Controlled, 2-Way, 4-Period Crossover Study To Assess Effects Of PF-02545920 On Ketamine-Induced Aberrant Prefrontal Response To Associative Learning In Healthy Subjects
Brief Title: Effects Of PF-02545920 On Ketamine-Induced Abnormal Prefrontal Brain Response To Associative Learning In Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: A8241014
Record Dates: First submitted 2010-11-05; First posted 2010-11-19 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: PF-02545920; ketamine; fMRI; associative Learning
MeSH Terms: interventions — Sodium Chloride; 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Saline/PF-02545920 (Experimental): Treatments are co-administered
  Interventions: Other: Saline; Drug: PF-02545920
- Ketamine/PF-02545920 (Experimental): Treatments are co-administered
  Interventions: Other: Ketamine; Drug: PF-02545920
- Saline/Placebo (Placebo Comparator): Treatments are co-administered
  Interventions: Other: Saline; Other: Placebo
- Ketamine/Placebo (Experimental): Treatments are co-administered
  Interventions: Other: Ketamine; Other: Placebo

INTERVENTIONS:
Other: Saline — Saline infusion for 56 minutes
  Arms: Saline/PF-02545920
Drug: PF-02545920 — PF-02545920 10 mg single dose
  Arms: Saline/PF-02545920
Other: Ketamine — Ketamine 0.23 mg/kg bolus over one min; and 0.58 mg/kg/hour maintenance for 56 minutes
  PF-02545920 10 mg tablet
  Arms: Ketamine/PF-02545920
Drug: PF-02545920 — PF-02545920 10 mg tablet single dose
  Arms: Ketamine/PF-02545920
Other: Saline — Saline infusion for 56 minutes
  Arms: Saline/Placebo
Other: Placebo — Placebo tablet single dose
  Arms: Saline/Placebo
Other: Ketamine — Ketamine 0.23 mg/kg bolus over one min; and 0.58 mg/kg/hour maintenance for 56 minutes
  Arms: Ketamine/Placebo
Other: Placebo — Placebo tablet single dose
  Arms: Ketamine/Placebo

SUMMARY:
To evaluate whether PF-02545920 reduces the effects of ketamine on brain activation during causal learning as measured by fMRI compared to placebo in healthy human subjects, and to evaluate whether behavioral measures of abnormal causal learning under ketamine are reduced by treatment with PF 02545920.

DETAILED DESCRIPTION:
The study was terminated on November 2, 2012 due to a reassessment of the likelihood of the study meeting its scientific objectives in light of data with the investigational drug obtained from another clinical study. The decision to terminate the trial was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 45 years, inclusive. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs). (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Right handed as determined by handedness questionnaire.
* Able to read and write English as a primary language.

Exclusion Criteria:

* Female subjects who are pregnant or breastfeeding.
* Any evidence of significant psychosis-like symptoms.
* Known sensitivity to ketamine.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2011-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Lateral prefrontal cortex activation as measured by functional MRI (fMRI) BOLD imaging during causal learning and working memory tasks | Day 1 of each treatment period

SECONDARY OUTCOMES:
Lateral prefrontal cortex activation during causal learning and working memory tasks as measured by arterial spin labelling imaging | Day 1 of each treatment period
Causal learning task prediction error score for stimulus/outcome associations across 3 stages of learning and expectancy violation | Day 1 of each treatment period
N-back working memory task number correct | Day 1 of each treatment period
Positive and Negative Syndrome Scale (PANSS) positive and negative subscale total score | Day 1 of each treatment period
Clinician administered dissociative states scale (CADSS) total score | Day 1 of each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8241014&StudyName=Effects%20Of%20PF-02545920%20On%20Ketamine-Induced%20Abnormal%20Prefrontal%20Brain%20Response%20To%20Associative%20Learning%20In%20Healthy%20Subjects%20